CLINICAL TRIAL: NCT05465031
Title: Sacubitril/Valsartan in PriMAry preventIoN of the Cardiotoxicity of Systematic breaST canceR trEAtMent
Brief Title: Sacubitril/Valsartan in PriMAry preventIoN of the Cardiotoxicity of Systematic breaST canceR trEAtMent (MAINSTREAM)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Silesian Centre for Heart Diseases (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LCZ696ABM001.001
Record Dates: First submitted 2022-07-04; First posted 2022-07-19 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Neoplasm, Breast; Breast Diseases; Antihypertensive Agents; Sacubitril/Valsartan; Angiotensin II Type 1 Receptor Blockers; Angiotensin Receptor Antagonists; Molecular Mechanisms of Pharmacological Action; Heart Failure; Cardiac Toxicity; Cancer, Therapy-Related; Cancer Therapy-Related Cardiac Dysfunction; Cardiotoxicity
Keywords: LCZ696; Sacubitril/Valsartan; Magnetic Resonance Imaging; Echocardiography; Cardio-oncology; Breast Cancer; Cardiotoxicity; Anthracyclines; Trastuzumab; Heart failure; Cardioprotection
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases; Heart Failure; Cardiotoxicity; Neoplasms, Second Primary | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Sacubitril/Valsartan (Experimental): After assessment of the tolerance of the drug during the single-blind period, during the which the starting dose of the drug of 100 mg b.i.d. should be increased after two weeks to the target dose 200 mg b.i.d, the patients will be randomized in 1:1 ratio to either intervention or placebo group. In the experimental arm, the patients after randomization will receive the dose 200 mg b.i.d of sacubitril/valsartan for the course of the study. If the patients does not tolerate the target dose of 200 mg b.i.d., the reduction of the drug dose to 100 mg b.i.d. will be possible at the discretion of the physician-in-charge.
  Interventions: Drug: Sacubitril-valsartan
- Placebo (Placebo Comparator): After assessment of the tolerance of the drug during the single-blind period, during the which the starting dose of the drug of 100 mg b.i.d. should be increased after two weeks to the target dose 200 mg b.i.d, the patients will be randomized in 1:1 ratio to either intervention or placebo group. In the placebo arm, the patients will receive the matching placebo with an identical strategy of dose reduction as in the intervention group, at the discretion of the physician-in-charge.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sacubitril-valsartan — Sacubitril/valsartan (Entresto®) administered in the target dose of 200 mg b.i.d. (97/103 mg of sacubitril and valsartan respectively) for the period of 24 months. In case of target dose intolerance, the physician-in-charge will be able to reduce the dose to 100 mg b.i.d. (49/51mg of sacubitril and valsartan respectively). Physicians will be strongly encouraged to evaluate the possibility of drug dose uptitration to the target dose of 200 mg b.i.d.
  Arms: Experimental: Sacubitril/Valsartan
Drug: Placebo — Placebo matching the sacubitril/valsartan (Entresto®) administered in the target dose matching the dosing of 200 mg b.i.d. (97/103 mg) for the period of 24 months. In case of intolerance of target dose of placebo, the physician-in-charge will be able to reduce the dose to placebo matching the dose of 100 mg b.i.d. (49/51mg). Physicians will be strongly encouraged to evaluate the possibility of drug dose uptitration to the target dose of placebo matching the dose of 200 mg b.i.d.
  Arms: Placebo

SUMMARY:
Breast cancer is the most commonly cancer in women in the overall global population. According to the World Cancer Research Fund International, there were more than 2.25 million new cases of breast cancer in women in 2020. Although the modern treatment strategies, based on the complex care, which consists of surgery, radiotherapy, hormone therapy, and targeted chemotherapy directed at specific cancer molecules have substantially reduced the risk of death due to breast cancer, their wide adoption results in the wider prevalence of cardiotoxicity, defined as either symptomatic heart failure, or asymptomatic contractile dysfunction. The occurrence of cardiotoxicity induced by anti-cancer therapies is estimated at 5-15%, and its development is the primary cause of therapy termination, which significantly reduces the probability of the efficacy of treatment. Several attempts have been made to determine the efficacious preventive strategy, which could diminish the risk of cancer-therapy induced cardiotoxicity. The results of the prior studies indicated a trend towards lower risk of troponin elevation, or left ventricular contractile dysfunction with the introduction of drugs interfering with the renin-angiotensin-aldosterone (RAA) axis, which constitute the primary treatment modality in heart failure with reduced ejection fraction (HFrEF). Sacubitril/valsartan, the novel therapeutic agent, has been demonstrated to significantly improve prognosis in patients with HFrEF. Prior retrospective, small, single-center studies have shown that treatment with sacubitril/valsartan may reduce the risk of cancer-therapy induced cardiotoxicity, or reverse contractile dysfunction caused by anti-cancer therapy. However, no large randomized data confirmed these findings.

Therefore, the Sacubitril/Valsartan in PriMAry preventIoN of the cardiotoxicity of systematic breaST canceR trEAtMent) study, has been designed to verify, whether the preventive use of sacubitril/valsartan administered in the doses recommended in patients with HFrEF in breast cancer patients undergoing adjuvant chemotherapy with anthracyclines or anthracyclines and HER-2 monoclonal antibodies, will reduce the incidence of cardiotoxicity defined as impaired left ventricular systolic function on transthoracic echocardiography (TTE). In the trial, a total of 480 patients with histologically confirmed breast cancer, who are eligible for chemotherapy with anthracyclines or anthracyclines and HER-2 monoclonal antibodies, will undergo 1:1 randomization to either preventive treatment with sacubitril/valsartan or placebo. The patients will be followed for 24 months, and will have repetitive efficacy and safety examinations, including echocardiography, MRI (optionally), electrocardiography including 24-h Holter monitoring, blood tests, functional capacity tests and quality of life assessment.

DETAILED DESCRIPTION:
MAINSTREAM is a prospective, multicentre, randomised, placebo-controlled, double-blind, parallel-group, investigator-initiated clinical trial. The study is powered to demonstrate the difference between the groups in the primary endpoint, which has been defined as the occurrence of a decrease in LVEF by ≥ 5% assessed by transthoracic echocardiography (TTE) within 24 months. Approximately 600 patients will be recruited in three tertiary supraregional Polish oncology centers. Of those patients, after an estimated dropout, during the single-blinded phase of drug uptitration to the target dose, 480 will be randomized in a 1:1 ratio into sacubitril/valsartan or matching placebo.

In brief, patients with histologically confirmed, and phenotypically assessed breast cancer at an early stage, defined as stages I-III and oligometastatic IV stage, with a radical treatment plan, which includes surgery and the post- and/or pre-operative systemic treatment, will be included in the study. The patients must be classified in the 0-2 classes of the Eastern Cooperative Oncology Group. In the baseline echocardiography analysis, the LVEF must be ≥50% and the patients must be in the sinus rhythm. The patients who underwent prior therapy with anthracyclines and/or left-sided radiotherapy, suffered from myocardial infarction within the preceding 3 months prior to the study, or have symptomatic, clinically relevant heart failure, will be excluded from the study. Similarly, patients with contraindications, or prone to the adverse effects of the studied drug, which includes patients with symptomatic hypotension, hyperkalemia defined as K+ higher than 5.5 mmol/L and estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 on the screening visit, will also be considered ineligible to participate in this trial. Patients must not have been on treatment with ACE-I/ARB/ARNI at least in the 36 hours prior to study enrollment. According to the ESC guidelines on cardio-oncology, the inclusion and exclusion criteria for the trial define the vast majority of the studied population in the low- or moderate risk of cancer therapy-related cardiac dysfunction (CTRCD), however, the inclusion of patients at high risk of either anthracycline- or anti-HER-2-associated CTRCD, such as patients aged ≥80 years, is not impossible. No very high-risk patients will be considered eligible for enrollment.

After assessment of the inclusion and exclusion criteria, and all examinations, including the echocardiography assessment, the patients will begin the single-blinded phase of treatment with sacubitril/valsartan during the screening visit. The MRI study may be performed according to the availability of the method in each participating facility. The initial dosing of the drug will be 49/51 mg twice daily, which should be uptitrated to the target dose of 97/103 mg twice daily at the Run-in-visit scheduled at 6-8 days from the initial evaluation and drug introduction, tolerance permitting. After further 6-8 days of single-blinded treatment with target dose of sacubitril/valsartan, providing satisfactory tolerance of the drug, the patients will undergo randomization at the Randomization visit.

Providing the patient signed informed consent, is fully eligible for randomization, and underwent the single-blinded study treatment regimen with satisfactory tolerance, the patient will be randomized with the use of an electronic, centralized randomization system, blinded to the patient's characteristics, to either interventional group, which will be administered with sacubitril/valsartan, or the placebo group. The system will dynamically randomly allocate patients to the two groups in a 1:1 ratio.

After randomization, the patients will follow treatment with either sacubitril/valsartan or a matching placebo, for a maximum of 24 months. During this period, three study visits are planned, at 3 months, 12 months, and 24 months from randomization. At each visit, the patients will be assessed for the medical presentation, undergo laboratory and imaging studies, and will be assessed for the presence of adverse events. In patients, who will be unable to tolerate the target dose of the study drug of 97/103 mg twice daily, the dose can be down-titrated to 49/51 mg twice daily at the investigator's discretion (after having considered whether there is any other concomitant medication that could act as a parallel contributor to the lower tolerance of the drug). If the dose of 49/51 mg twice daily cannot be tolerated, the dose could be temporarily lowered by half for a period of two weeks. However, if after that period the uptitration of the dose is impossible, the patients will have to be excluded from further participation in the trial. The physicians will be strongly encouraged to foster the continuation of the target dose of the study drug, based on their assessment of the patient's condition.

The primary endpoint of the study has been defined as the occurrence of a reduction in LVEF by ≥ 5% assessed by TTE within 24 months. Among the secondary endpoints of the study, the clinical composite endpoint of death from any cause or hospitalization for heart failure and its components will be analysed, as well as the wide spectrum of echocardiographic, electrocardiographic, laboratory, and clinical outcomes, including the CTRCD resulting in the need to implement treatment consistent with the ESC guidelines on cardio-oncology. To maintain utmost objectivity, all examinations performed in relation to the study, including the echocardiographic, electrocardiographic, and magnetic resonance imaging analyses will be sent using 3D option ImageCom (TOMTEC Imaging Systems GmbH, Germany) - a multi-modality, vendor-neutral 3D/4D viewer - to the core laboratory where their results will be analysed by two independent investigators blinded to the patient's randomization status.

Breast cancer treatment The patients should be treated according to the standard protocols of the participating centres, with the intention of radical treatment based on the surgical excision of cancer, with addition of either pre- or post-surgical chemo- and/or radiotherapy. The choice of the scheme of oncological treatment will be at the discretion of the treating oncologist and will be performed after analysis of the risk of recurrence, the potential response to a particular type of treatment, with consideration of possible drug-related adverse effects, and patient's co-morbidities and preferences. All decisions, including the scheme of therapy, will be performed in accordance with the recommendations of the Polish Society of Clinical Oncology.

Pre-operative and post-operative chemotherapy with alkylating drugs, which include anthracyclines, usually in multi-drug regimens, will begin most commonly, with the initiation of anthracyclines (4 cycles or 3 cycles of EC). In routine perioperative treatment, trastuzumab will be administered̨ for 12 months, but shorter regimens (6 months) may be considered in individual situations, however, due to the cardiotoxic effects of trastuzumab, it will not be routinely given concomitantly with anthracyclines.

As there are currently no data regarding the potential differences in the pharmacodynamics and pharmacokinetics, and consequently efficacy and safety of sacubitril/valsartan prophylactic treatment in patients with breast cancer and systemic therapy, there may be genetic biomarkers defining the disease susceptibility and prognosis, as well as the response to treatment. For each patient who gives informed consent to participate in the study, an additional blood sample will be taken at the first visit. After completion of the study, the subanalysis of the trial will be attempted based on the genetic profile aiming at defining the genetic pattern characterizing the response to sacubitril/valsartan for the prevention of cardiotoxicity caused by anthracyclines and/or anti-HER-2 targeted drugs.

At the screening visit and completion of the study, the patient will undergo TTE, which according to the recent ESC Guidelines on cardio-oncology has been defined as the first-line modality in assessment of cardiac function in oncological patients. The assessment of LVEF with the use of 3D echocardiography will be preferred in all patients, although in selected cases a two-dimensional LVEF assessment will be accepted. In every patient, the assessment of global longitudinal strain will be recommended. The investigator performing the echocardiography will be blinded to the patient's randomization scheme. All images will be sent to the core laboratory. The quality of life will be assessed with the 36-Item Short Form Survey (SF-36) questionnaire at the screening visit and at the completion of the study.

Laboratory tests The details of the blood tests performed during each study visit are presented in Table 4. All blood samples will be performed at fasting, on the day of the study visits, and analysed in the local laboratories of the three participating oncology centres. The blood sample for genetic testing in patients who sign an additional consent for genetic evaluation will be collected only on the screening visit and stored locally for the eventual transfer into the biobank of the Maria Sklodowska-Curie Institute - Oncology Centre (MSCI), Gliwice, Poland for further analyses. High-sensitivity cardiac troponin (with a preference to measure cardiac troponin T over troponin I due to previously described variability in the results of the latter), as well as N-terminal prohormone of brain natriuretic peptide (NT-proBNP), will be assessed using assays at the local laboratories of the participating oncology centres during study visits and at any time when deemed necessary by the physician-in-charge, or as supported by the local treatment protocols established by the participating centres and with reference to the ESC guidelines on cardio-oncology. The investigators will be blinded to the patients' randomization results.

Intervention in case of HF development Based on the prior studies, it is estimated that approximately 20% of patients from the placebo arm and 10% of study drug arm might develop a certain degree of cardiotoxicity and require introduction of cardioprotective agents. The diagnosis of CTRCD should be based on the assessment of TTE and/or high-sensitivity cardiac troponin, as well as NT-proBNP. The intervention in case of development of either symptomatic, or asymptomatic CTRCD should be in line with current ESC guidelines on cardio-oncology and may include discontinuation or temporary interruption of chemotherapy, or continuation of treatment with thorough patient monitoring, while the study drug/placebo might be terminated or continued, depending on the severity of CTRCD.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Female gender, aged 18 years and over
* Patients with histologically confirmed breast cancer and complete assessment of tumor phenotype (Estrogen receptor - ER, Progesterone receptor - PR, Human epidermal growth factor receptor 2 - HER2, Kiel - Ki67)
* Ability to take oral medication and willingness to adhere to the planned regimen
* Tumor grade IA-IIIC or oligometastatic grade IV
* Radical treatment plan including surgery
* Plan of use of systemic treatment (preoperative, postoperative or combined) with anthracyclines and/or anti-HER2 drugs
* Eastern Cooperative Oncology Group (ECOG) 0-2 general status
* LVEF ≥ 50% as assessed by echocardiography
* Sinus rhythm

Exclusion Criteria:

* Prior anthracycline-based chemotherapy and/or thoracic radiotherapy (prior to diagnosis of the cancer being the present cause of therapy)
* Clinically relevant HF (NYHA II-IV)
* Myocardial infarction (MI) within the last < 3 months
* Symptomatic hypotension or systolic blood pressure (SBP) < 90 mmHg
* Significant valvular disease, symptomatic coronary artery disease (CCS>2), significant atrioventricular (AV) block, symptomatic sinus node dysfunction
* Expected survival <12 months
* Glomerular filtration rate (GFR) <30 ml/min/1.73 m2 (screening visit)
* K+>5.5mmol/L (screening visit)
* Contraindications to angiotensin converting enzyme inhibitor (ACE-I)/angiotensin II receptor blocker (ARB) or LCZ696 if not listed among criteria
* Active untreated liver disease
* Pregnancy
* Conditions/circumstances that may lead to non-compliance with medical staff recommendations (e.g. active drug/alcohol dependence, poorly controlled mental illness)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — As breast cancer is primarily the female malignancy, the studied population will be limited to female patients
Enrollment: 600 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction (LVEF) by ≥5% | Within 24 months from the randomization visit
  Reduction of LVEF assessed on transthoracic echocardiography (TTE)

SECONDARY OUTCOMES:
Death from any cause or hospitalization for heart failure | From Randomization till the end of blinded therapy - at 24 months
  Composite clinical endpoint
Death from any cause | From Randomization till the end of blinded therapy - at 24 months
  Clinical endpoint
Death from cardiovascular causes | From Randomization till the end of blinded therapy - at 24 months
  Clinical endpoint
Hospitalization for other cardiovascular causes | From Randomization till the end of blinded therapy - at 24 months
  Clinical endpoint
Change in left ventricular ejection fraction by ≥ 5% | From Randomization till the end of blinded therapy - within 24 months
  Reduction of LVEF assessed on magnetic resonance imaging (MRI)
Occurrence of diastolic dysfunction (TTE) within 24 months of randomization | From Randomization till the end of blinded therapy - at 24 months
  Diastolic dysfunction assessed on echocardiography
- Development of pathological pericardial fluid volume or increase in pericardial fluid volume from baseline | From Randomization till the end of blinded therapy - at 24 months
  Assessed with any available clinical modality
Occurrence of cardiac tamponade | From Randomization till the end of blinded therapy - at 24 months
  Assessed with any clinical modality
Occurrence of pericarditis | From Randomization till the end of blinded therapy - at 24 months
  Assessed with any clinical modality
Occurrence of myocarditis | From Randomization till the end of blinded therapy - at 24 months
  Assessed with any clinical modality
Development of ventricular arrhythmias | From Randomization till the end of blinded therapy - at 24 months
  Assessed with any clinical modality
Development of supraventricular arrhythmias | From Randomization till the end of blinded therapy - at 24 months
  Assessed with any clinical modality
Presence of conduction disturbances | From Randomization till the end of blinded therapy - at 24 months
  Assessed with any clinical modality
Changes in corrected QT interval | From Randomization till the end of blinded therapy - at 24 months
Changes in B-type natriuretic peptide (BNP) or N-terminal prohormone of brain natriuretic peptide (NT pro-BNP) (pg/mL) | From Randomization till the end of blinded therapy - at 24 months
  Assessed with serial laboratory measurements
Changes in cardiac troponins (cardiac troponin T preferred over troponin I) (ng/L) | From Randomization till the end of blinded therapy - at 24 months
  Assessed with serial laboratory measurements

CONTACTS AND LOCATIONS:
Overall Officials: Mateusz Tajstra, Principal Investigator — 3rd Department of Cardiology, School of Medical Sciences in Zabrze, Medical University of Silesia, Katowice; Silesian Center for Heart Diseases
Locations (4):
- Poland (4):
  - Regional Cancer Centre in Opole, Opole, Opole Voivodeship
  - Maria Sklodowska-Curie Institute - Oncology Centre (MSCI), Gliwice Branch, Gliwice, Silesian Voivodeship
  - Silesian Center for Heart Diseases, Zabrze, Silesian Voivodeship
  - Holy Cross Cancer Centre, Cardio-Oncology Division, Kielce, Świętokrzyskie Voivodeship

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tajstra M, Dyrbus M, Rutkowski T, Skladowski K, Sosnowska-Pasiarska B, Gozdz S, Radecka B, Staszewski M, Majsnerowska A, Myrda K, Nowowiejska-Wiewiora A, Skoczylas I, Rymkiewicz I, Niklewski T, Nowak J, Przybylowski P, Gasior M, Jarzab M. Sacubitril/valsartan for cardioprotection in breast cancer (MAINSTREAM): design and rationale of the randomized trial. ESC Heart Fail. 2023 Oct;10(5):3174-3183. doi: 10.1002/ehf2.14466. Epub 2023 Jul 14. PMID 37449716